CLINICAL TRIAL: NCT03974269
Title: Hypnosis Versus Intravenous Sedation With Concentration Objective (SIVOC) by Remifentanil During TAVI Procedures: Impact on Perioperative Confusion
Brief Title: Hypnosis Versus SIVOC by Remifentanil During TAVI Procedures : Iloact on Peripoperative Confusion
Acronym: HYPSED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018-A00563-52
Record Dates: First submitted 2019-04-23; First posted 2019-06-04 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Confusion
Keywords: Hypnosis; Delirium; Transcatheter aortic valve implantation
MeSH Terms: conditions — Confusion; Delirium

STUDY DESIGN:
Intervention Model Description: 2 arms : hypnosis group and sedation group
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis arm (Active Comparator): TAVI procedures will be either Medtronic Corevalve, or Edwards Sapien implantations, at operator's discretion. All procedures will be supervised by one of the two senior interventional cardiologists. Hypnosis sessions will be performed by two trained anesthesiologists, and Remifentanil sedations will be administered by the rest of the anesthesiologists staff. Postoperative care will be provided in the CICU for the 3 first postoperative days at least.
  Interventions: Procedure: TAVI : Transcatether Aortic Valve Implantation
- Sedation arm (Placebo Comparator): TAVI procedures will be either Medtronic Corevalve, or Edwards Sapien implantations, at operator's discretion. All procedures will be supervised by one of the two senior interventional cardiologists. Hypnosis sessions will be performed by two trained anesthesiologists, and Remifentanil sedations will be administered by the rest of the anesthesiologists staff. Postoperative care will be provided in the CICU for the 3 first postoperative days at least.
  Interventions: Procedure: TAVI : Transcatether Aortic Valve Implantation

INTERVENTIONS:
Procedure: TAVI : Transcatether Aortic Valve Implantation — TAVI procedures will be either Medtronic Corevalve, or Edwards Sapien implantations, at operator's discretion. All procedures will be supervised by one of the two senior interventional cardiologists. Hypnosis sessions will be performed by two trained anesthesiologists, and Remifentanil sedations will be administered by the rest of the anesthesiologists staff. Postoperative care will be provided in the CICU for the 3 first postoperative days at least.

SUMMARY:
TAVI has become a credible alternative to conventional cardiac surgery in aged high-risk patients with aortic valve stenosis. A large part of these procedures are performed with sedation using remifentanil target-controlled infusion plus local anesthesia. However, a significant proportion of the patients experience postoperative delirium, with subsequent worsened outcomes, time-consuming interventions, and increased costs. The use of hypnosis before and during TAVI could decrease the incidence of postoperative delirium thanks to less opioids and hypnotics consumption. Thus, the investigators ought to evaluate the potential advantages of hypnosis vs. remifentanil target controlled-infusion during TAVI procedures.

DETAILED DESCRIPTION:
Each included patient will randomly be assigned either to the hypnosis group or to the remifentanil group. Patients of the hypnosis group will have one preoperative and one perioperative hypnosis session with a qualified anesthesiologist. Patients of the remifentanil group will receive sedation with remifentanil, administered using a pre specified target controlled-infusion protocol.

Incidence of delirium will be recorded in the cardiac intensive care unit (CICU) during the first 72 postoperative hours, using the Confusion Assessment Method in the ICU (CAM-ICU). Incidence of other complications such as episodes of oxygen desaturation, vascular wound, stroke, general anesthesia requirement and inhospital death will be recorded, as well as procedure duration, hospital length of stay, patient satisfaction and operator comfort.

Transcatheter aortic valve implantation (TAVI) procedures are frequently complicated with postoperative delirium.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring transfemoral approach TAVI without general anesthesia
* For adult patients : age greater than or equal to 18 years
* Patients affiliated to a social security scheme

Exclusion Criteria:

* Patient whose age is less than 18 years
* Approach with general anesthesia
* Patient not responding to Hypnosis: unmotivated, non-cooperating, not confident
* Other than transfemoral approach : carotid, trans-apical or sternotomy or thoracotomy procedure
* chronic psychosis, bilateral deafness without hearing aids,
* emergency procedure,
* inability to communicate (severe dementia, non-French speaker),
* declined participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2018-06-11 (Actual); Primary Completion 2020-06-11 (Estimated); Study Completion 2021-06-11 (Estimated)

PRIMARY OUTCOMES:
Occurrence of a postoperative delirium episode | 72 hours
  Assessment of the level of postoperative confusion will be measured at the CAM-ICU (Confusion Assessment Method Intensive Care Unit) scale. The CAM-ICU scale is a questionnaire based on 4 items. The diagnosis of delirium requires the presence of 3 of the 4 criteria. Criteria 1 and 2 are still required, with criteria 3 or 4.

SECONDARY OUTCOMES:
Incidence of intraoperative complications | 72 hours
  Intraoperative complications

OTHER OUTCOMES:
Length of the procedures | 72 hours
  Duration of the procedure in the catheterization room.
Comfort felt by the patient | 72 hours
  visual scale : score from 0 to 4: 0 not comfortable at all, 4 very
Operator comfort | 72 hours
  visual scale : score from 0 to 10: 0 bad conditions, 10 excellent conditions
Anxiety assessment | 72 hours
  visual scale : score from 0 to 10: 0 no anxiety, 10 worst possible anxiety
Patient pain | 72 hours
  visual scale : score from 0 to 10: 0 no pain, 10 maximum pain imaginable
episodes of nausea and vomiting at the 1st meal after the procedure | 72 hours
  Number of episodes of nausea and vomiting at the 1st meal after the procedure
Patient satisfaction at the end of the procedure | 72 hours
  visual scale : score from 0 to 10: 0 not at all satisfied, 10 very satisfied
Incidence of anesthetic procedure in both groups: | 72 hours
  Number of anesthetic procedure failures in both groups
  * in the group Hypothesis defined by a transition to a SIVOC sedation or a general anesthesia.
  * In the Sedation group defined by a transition to "hypnosis" or "hypnotic accompaniment" or general anesthesia
Average lengths of stay, | 72 hours
  Total length of stay in the patient's hospital
Incidence of mortality during the hospital stay | 72 hours
  Occurrence of a death during the hospital stay
Costs of hospital stays. | 72 hours
  Evaluation of the costs of hospital stays.

CONTACTS AND LOCATIONS:
Overall Officials: Marina Rubatti, Principal Investigator — Hôpital Marie Lannelongue
Locations (1):
- Hopital Marie Lannelongue, Le Plessis-Robinson, France

IPD SHARING:
Plan to Share IPD: No